CLINICAL TRIAL: NCT03644147
Title: Additive Effect of Intravenous Acetaminophen Administered at the End of Surgery on Postoperative Pain Control With Nefopam and Fentanyl-based Patient-controlled Analgesia: A Double-blind Randomized Controlled Trial
Brief Title: Additive Effect of Intravenous Acetaminophen on Postoperative Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1807-151-961
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Gynecologic Disease
MeSH Terms: conditions — Pain, Postoperative; Genital Diseases, Female | interventions — Acetaminophen; Therapeutics

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients in this group will receive 1 gram of acetaminophen intravenously after the end of surgery.
  Interventions: Drug: Acetaminophen
- Control (No Intervention): Patients in this group will receive 100 ml of normal saline intravenously after the end of surgery.

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen will be intravenously administrated to treatment group after the end of surgery.
  Other Names: treatment
  Arms: Treatment

SUMMARY:
This study aimed to evaluate the additive effect of acetaminophen on postoperative pain control in patients receiving nefopam and fentanyl-based patient-controlled analgesia.

Participants undergoing laparoscopic hysterectomy will be randomly assigned to treatment group or control group. After end of surgery, acetaminophen or normal saline (placebo) will be administered intravenously depending on the group assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total laparoscopic hysterectomy due to uterine myoma, cervical cancer, endometriosis, uterine prolapse

Exclusion Criteria:

* Liver disease (aspartate transaminase OR alanine transaminase > 80 IU/L)
* Chronic kidney disease (GFR < 30 ml/min/1.73m2)
* History of drug allergy
* Chronic pain lasting more than 3 months
* Conversion to laparotomy
* Complex surgery (co-operation with colon surgeon or urologist)
* Limitation in expressing pain

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Total volume of administered analgesics during postoperative 24 hours | 24 hours
  morphine equivalent dose of patient-controlled analgesics administered during first 24 hours after end of surgery

SECONDARY OUTCOMES:
Pain score | 24 hours
  11-point numeric rating scale ranging from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Patient satisfaction score | 24 hours
  11-point numeric rating scale ranging from '0' representing one extreme (e.g. "extremely dissatisfied") to '10' representing the other extreme (e.g. "extremely satisfied")
Postoperative nausea and vomiting | 24 hours
  4-scales scoring (none; mild; moderate; severe)
Opioid-related adverse effect | 24 hours
  Incidence of respiratory, gastrointestinal, and central nervous system complications
Use of alternative analgesics | 24 hours
  Additional administration of other analgesics
Length of stay | From date of hospital admission until the date of discharge, an average of 1 week
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Pf., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Nam S, Yoo S, Park SK, Kim JT. Additive effect of a single intravenous dose of acetaminophen administered at the end of laparoscopic hysterectomy on postoperative pain control with nefopam and fentanyl-based patient-controlled analgesia: a double-blind, randomized controlled trial. BMC Anesthesiol. 2025 Feb 20;25(1):88. doi: 10.1186/s12871-025-02971-w. PMID 39979845